CLINICAL TRIAL: NCT03051776
Title: Kinesio Taping Versus Compression Garments in the Treatment of Breast Cancer-Related Lymphedema. Randomized Crossover Trial.
Brief Title: Kinesio Taping Versus Compression Garments for Breast Cancer-Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Violeta Pajero Otero (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other); University of Castilla-La Mancha (Other)
Responsible Party: Sponsor-Investigator, Violeta Pajero Otero, Physiotherapist at the Mammary Pathology Unit, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: InveCuidRhKM
Record Dates: First submitted 2017-02-08; First posted 2017-02-14 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer Lymphedema
Keywords: Compression garments; Kinesio Taping; Breast Cancer-Related Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: Two treatmet phases, with a four week wash out period bewtween them:
  * A four week phase with Kinesio Taping
  * A four week phase with compression garments.
Who Masked: Outcomes Assessor
Masking Description: The statistical analysis will be supervised by staff of the Scientific Support Unit: Epidemiology and Biostatistics (i+12), Hospital Universitario 12 de Octubre with the variables coded to blind the analyst.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping (Experimental): It was done a four week phase with Kinesio Taping in the arm affected with lymphedema.
  Interventions: Other: Kinesio Taping
- Compression garment (Active Comparator): It was done a four week phase with Compression garment in the arm affected with lymphedema.
  Interventions: Other: Compression Garment

INTERVENTIONS:
Other: Kinesio Taping
  Arms: Kinesio Taping
Other: Compression Garment
  Arms: Compression garment

SUMMARY:
Breast cancer-related lymphedema (BCRL) tends to become chronic and progressive. Current therapies have modest results for this condition. Compression garments (CG) prevent the worsening of lymphedema and even improve it, during periods between treatments of physical therapy. Kinesio Taping(KT) is being recently used for lymphedema, although little evidence backs it. The aim of this study is to compare the reduction of lymphedema volume with both therapies.

DETAILED DESCRIPTION:
Primary end points: to evaluate whether the decrease in BCRL volume is different for a 4-week treatment with KT than with CG.

Research design:

Randomized quasi-experimental clinical pilot study: initial sample randomly balanced into two groups . The initial sample was selected among the patients of "Breast Pathology Rehabilitation" at Hospital Universitario 12 de Octubre . The planned sample size was 30.

Cross Design: it made possible to evaluate two different treatments in the same patient, cancelling intragroup variability.

Open design: it was impossible to blind patients and physiotherapist researcher because of patent visual differences between the two therapies, CG or KT, both during application and while being worn, and even in the hours after its removal, due to the marks left on the skin. However, at least one external evaluator suitably trained was implemented and performed the randomisation of the groups and collected all patient data. Statistical study was also made by others (staff of the "Clinique Investigation Unit (i+12)" of Hospital Universitario 12 de Octubre) with coded variables to blind the analyst.

ELIGIBILITY:
Inclusion Criteria:

1. Suffering from clinically significant breast cancer-related lymphedema at least since three months ago.
2. Having a Compression Garment suitable for the lymphedema arm

Exclusion Criteria:

1. Physiotherapy treatment for lymphedema during the 4 weeks before study start (pre-wash phase).
2. Metastasis breast cancer or other tumour.
3. Treated with systemic chemotherapy and /or radiotherapy at that time
4. Heart Failure or Renal Failure.
5. Using Diuretics.
6. Bilateral axillary lymphadenectomy.
7. Cognitive impairment or delay that impedes understanding the study's instructions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-03 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-03-30 (Actual)

PRIMARY OUTCOMES:
Estimated volumen of the upper limb. | Four weeks during each treatment phase
  Truncated Cone Formula.

SECONDARY OUTCOMES:
Symptoms associated with BCRL (pain, heaviness, pressure and hardness) using modified visual analogue scale (VAS). | Four weeks during each treatment phase
  Wong-Baker faces pain rating scale.
Goniometry of Upper Limb. | Four weeks during each treatment phase
  Goniometry of shoulder, elbow, wrist and hand.

CONTACTS AND LOCATIONS:
Overall Officials: Violeta Pajero Otero, MRes, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No